CLINICAL TRIAL: NCT03138629
Title: Expanded Access to VAL-083
Status: No longer available | Type: Expanded Access
Sponsor: Kintara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DLM-17-002
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: VAL-083 — VAL-083 will be administered intravenously

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to VAL-083 (dianhydrogalactitol) prior to approval by the local regulatory agency. Availability will depend on territory eligibility. Participating sites will be added as they apply for and are approved for the EAP. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patient has relapsed/refractory disease and exhausted all standard treatments.

Exclusion Criteria:

* Patient is eligible for a VAL-083 clinical trial.
* Patient has previously received VAL-083 for the same disease.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult